CLINICAL TRIAL: NCT04148989
Title: Effects of Code Sepsis Implementation on Emergency Department (ED) Sepsis Care
Acronym: Code Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Ithan Peltan, Clinical Investigator, Intermountain Health Care, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1051053; K23GM129661 (NIH)
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
Keywords: Sepsis; Clinical Protocols; Emergency Medicine
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Patients presenting to the intervention emergency department after implementation of the care reorganization intervention - "Code Sepsis protocol" - will be compared to patients presenting prior to the intervention. Patients presenting to control emergency departments will receive usual care both before and after Code Sepsis implementation and are included in this study to control for changes in intervention-site outcomes over time unrelated to the tested intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-implementation usual care (intervention site) (No Intervention): Adult patients age ≥18 years who receive usual care after presenting to the ED of the intervention hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation). The primary analysis will focus on the subset of patients with sepsis.
- Code Sepsis post-implementation (intervention site) (Experimental): Adult patients age ≥18 years presenting to the ED of the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation). The primary analysis will focus on the subset of patients with sepsis.
  Interventions: Other: Code Sepsis protocol (full implementation)
- Pre-implementation usual care (control sites) (No Intervention): Adult patients age ≥18 years who receive usual care after presenting to the ED of the control hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital. The primary analysis will focus on the subset of patients with sepsis.
- Post-implementation usual care (control sites) (No Intervention): Adult patients age ≥18 years who receive usual care after presenting to the ED of the control hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital. The primary analysis will focus on the subset of patients with sepsis.

INTERVENTIONS:
Other: Code Sepsis protocol (full implementation) — Implementation of a coordinated, structured, multidisciplinary team-based protocol for initial evaluation and treatment of ED patients with suspected sepsis.
  Arms: Code Sepsis post-implementation (intervention site)

SUMMARY:
Sepsis is a life-threatening complication of infection that can be difficult to recognize and treat promptly. Timely administration of antibiotics for emergency department (ED) patients with sepsis is challenging. The goal of this study is to determine the potential effectiveness and unintended consequences of reorganizing ED care for patients with suspected sepsis.

ELIGIBILITY:
Inclusion criteria (overall):

1. Adult (age ≥18 years)
2. ED patient at Intermountain Medical Center, Utah Valley Hospital, Dixie Regional Medical Center
3. Arrival to study emergency department (ED) during study period of 11/13/2018 to 2/12/2021.

Exclusion criteria (overall):

(1) Trauma patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180402 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ithan Peltan, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Hospital, Provo, Utah
  - Dixie Regional Medical Center, St. George, Utah

IPD SHARING:
Plan to Share IPD: Yes
In order to protect patient privacy and comply with relevant regulations, identified data will be unavailable. Requests for deidentified data from qualified researchers with appropriate ethics board approvals and relevant data use agreements will be processed by the Intermountain Office of Research, officeofresearch@imail.org.

REFERENCES:
- [Derived] Peltan ID, Bledsoe JR, Jacobs JR, Groat D, Klippel C, Adamson M, Hooper GA, Tinker NJ, Foster RA, Stenehjem EA, Moores Todd TD, Balls A, Avery J, Brunson G, Jones J, Bair J, Dorais A, Samore MH, Hough CL, Brown SM. Effectiveness and Safety of an Emergency Department Code Sepsis Protocol: A Pragmatic Clinical Trial. Ann Am Thorac Soc. 2024 Nov;21(11):1560-1571. doi: 10.1513/AnnalsATS.202403-286OC. PMID 38996086

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Hospitals
Groups:
- Pre-implementation Usual Care (Intervention Site): Adult patients age ≥18 years who received usual care after presenting with sepsis to the intervention hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation).
- Code Sepsis Post-implementation (Intervention Site): Adult patients age ≥18 years exposed to the intervention after presenting to the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation).
  Code Sepsis protocol (full implementation): Implementation of a coordinated, structured, multidisciplinary team-based protocol for initial evaluation and treatment of ED patients with suspected sepsis.
- Pre-implementation Usual Care (Control Sites): Adult patients age ≥18 years who received usual care after presenting to the control hospital emergency department with sepsis before implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
- Post-implementation Usual Care (Control Sites): Adult patients age ≥18 years who receive usual care after presenting to the control hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
Period: Pre-implmentation Period
Arm/Group | Pre-implementation Usual Care (Intervention Site) | Code Sepsis Post-implementation (Intervention Site) | Pre-implementation Usual Care (Control Sites) | Post-implementation Usual Care (Control Sites)
Started | 50437; 1 Hospitals | 0; 0 Hospitals | 56192; 2 Hospitals | 0; 0 Hospitals
Completed | 50437; 1 Hospitals | 0; 0 Hospitals | 56192; 2 Hospitals | 0; 0 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals
Period: Post-implmementation Period
Arm/Group | Pre-implementation Usual Care (Intervention Site) | Code Sepsis Post-implementation (Intervention Site) | Pre-implementation Usual Care (Control Sites) | Post-implementation Usual Care (Control Sites)
Started | 0; 0 Hospitals | 33415; 1 Hospitals | 0; 0 Hospitals | 40358; 2 Hospitals
Completed | 0; 0 Hospitals | 33415; 1 Hospitals | 0; 0 Hospitals | 40358; 2 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Groups:
- Code Sepsis Post-implementation (Intervention Site): Adult patients age ≥18 years presenting to the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation).
  Code Sepsis protocol (full implementation): Implementation of a coordinated, structured, multidisciplinary team-based protocol for initial evaluation and treatment of ED patients with suspected sepsis.
- Total: Total of all reporting groups
Arm/Group | Pre-implementation Usual Care (Intervention Site) | Code Sepsis Post-implementation (Intervention Site) | Pre-implementation Usual Care (Control Sites) | Post-implementation Usual Care (Control Sites) | Total
Number analyzed (Participants) | 50437 | 33415 | 56192 | 40358 | 180402
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [31 to 64] | 45 [31 to 63] | 49 [30 to 69] | 47 [29 to 68] | 47 [30 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27762 | 17177 | 30458 | 20624 | 96021
  Male | 22675 | 16238 | 25734 | 19734 | 84381
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8710 | 6354 | 6189 | 5176 | 26429
  Not Hispanic or Latino | 40120 | 25458 | 48753 | 33541 | 147872
  Unknown or Not Reported | 1607 | 1603 | 1250 | 1641 | 6101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 660 | 418 | 771 | 567 | 2416
  Asian | 1012 | 802 | 475 | 362 | 2651
  Native Hawaiian or Other Pacific Islander | 1802 | 1099 | 895 | 703 | 4499
  Black or African American | 1456 | 951 | 704 | 471 | 3582
  White | 41684 | 26964 | 51444 | 36003 | 156095
  More than one race | 110 | 112 | 115 | 111 | 448
  Unknown or Not Reported | 3713 | 3069 | 1788 | 2141 | 10711
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50437 | 33415 | 56192 | 40358 | 180402

OUTCOME MEASURES:

1. Primary Outcome: Door-to-antibiotic Time
Description: Time from sepsis patients' emergency department arrival to intravenous (or equivalent) antibiotic initiation
Time Frame: Up to 24 hours from ED arrival (an average of 3 hours)
Population: Restricted to participants who met sepsis criteria (acute organ failure plus suspected or confirmed infection) before ED departure.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Pre-implementation Usual Care (Intervention Site) - Sepsis Patients: Adult patients age ≥18 years who received usual care after presenting with sepsis to the intervention hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation).
- Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients: Adult patients age ≥18 years presenting with sepsis to the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation).
  Code Sepsis protocol (full implementation): Implementation of a coordinated, structured, multidisciplinary team-based protocol for initial evaluation and treatment of ED patients with suspected sepsis.
- Pre-implementation Usual Care (Control Sites) - Sepsis Patients: Adult patients age ≥18 years who received usual care after presenting with sepsis to the control hospital emergency department with sepsis before implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
- Post-implementation Usual Care (Control Sites) - Sepsis Patients: Adult patients age ≥18 years who receive usual care after presenting with sepsis to the control hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
minutes | 160 [114 to 219] | 146 [102 to 205] | 139 [102 to 176] | 140 [105 to 177]
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; Differences-in-differences analysis using multivariable gamma regression to estimate the change in outcome after versus before intervention implementation at the intervention site adjusted for the change observed at control sites and for subjects' age, sex, Elixhauser Comorbidity Score, ED arrival via ambulance, English language preference, temperature, systolic blood pressure, Acute Physiology Score, Sequential Organ Failure Assessment score, and ED-diagnosed source of infection; Test type: Superiority; p < 0.001, Regression, gamma; Mean Difference (Final Values) = -12.8, 95% CI 2-sided [-18.6 to -7.0] — Change in emergency department door-to-antibiotic time (minutes) associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

2. Secondary Outcome: All-cause 30-day Mortality
Description: Sepsis patient death on or before the 30th day after ED arrival
Time Frame: 30 days after ED arrival
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
Participants | 201 | 262 | 280 | 332
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; Differences-in-differences analysis using multivariable logistic regression to estimate the change in outcome after versus before intervention implementation at the intervention site adjusted for the change observed at control sites and for subjects' age, sex, Elixhauser Comorbidity Score, ED arrival via ambulance, English language preference, temperature, systolic blood pressure, Acute Physiology Score, Sequential Organ Failure Assessment score, and ED-diagnosed source of infection; Test type: Superiority; p = 0.45, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.68 to 1.19] — Change in all-cause 30-day mortality risk associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

3. Secondary Outcome: All-cause 1-year Mortality
Description: Sepsis patient death on or before the 365th day after ED arrival
Time Frame: 1 year after ED arrival
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
Participants | 467 | 483 | 603 | 628
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.10, Regression, Logistic; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.67 to 1.04] — Change in all-cause 1-year mortality risk associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

4. Secondary Outcome: All-cause In-hospital Mortality
Description: Sepsis patient death prior to hospital discharge
Time Frame: From the time of admission to hospital discharge (up to 1 year, average 14 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
Participants | 113 | 148 | 149 | 190
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.15, Regression, Logistic; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.53 to 1.10]; Change in all-cause in-hospital mortality risk associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

5. Secondary Outcome: Hospital Charges
Description: Amount charged to sepsis patient for their medical care during index ED visit and associated hospitalization
Time Frame: From the time of admission to hospital discharge (up to 1 year, average 14 days)
Population: Restricted to participants who met sepsis criteria (acute organ failure plus suspected or confirmed infection) before ED departure. Subjects who met sepsis criteria but were missing outcome data (N=80 overall) were also excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: US dollars * 1000
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2366 | 2061 | 2952 | 2692
US dollars * 1000 | 7.3 [3.6 to 14.3] | 15.0 [7.0 to 32.7] | 7.6 [3.8 to 14.7] | 15.2 [7.6 to 30.1]
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.71, Regression, gamma; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.4 to 2.1] — Change in hospital charges ($1000s) associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

6. Secondary Outcome: Hospital Length of Stay
Description: Length of time from sepsis patients' ED arrival until hospital discharge
Time Frame: From the time of admission to hospital discharge (up to 1 year, average 14 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
days | 2.7 [1.0 to 5.0] | 3.0 [1.1 to 6.1] | 2.7 [1.1 to 4.8] | 2.9 [1.2 to 5.6]
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.19, Regression, gamma; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1] — Change in hospital length of stay (days) associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

7. Other Pre Specified Outcome: Antibiotic Utilization'
Description: Fraction of all ED patients receiving antibiotics within 24 hours of ED arrival
Time Frame: Up to 24 hours from ED arrival (an average of 6 hours)
Measure: Count of Participants; unit: Participants
Groups:
- Pre-implementation Usual Care (Intervention Site) - All ED Patients: Adult patients age ≥18 years who receive usual care after presenting to the ED of the intervention hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation).
- Code Sepsis Post-implementation (Intervention Site) - All ED Patients: Adult patients age ≥18 years presenting to the ED of the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation).
- Pre-implementation Usual Care (Control Sites) - All ED Patients: Adult patients age ≥18 years who receive usual care after presenting to the ED of the control hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
- Post-implementation Usual Care (Control Sites) - All ED Patients: Adult patients age ≥18 years who receive usual care after presenting to the ED of the control hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
Arm/Group | Pre-implementation Usual Care (Intervention Site) - All ED Patients | Code Sepsis Post-implementation (Intervention Site) - All ED Patients | Pre-implementation Usual Care (Control Sites) - All ED Patients | Post-implementation Usual Care (Control Sites) - All ED Patients
Number analyzed (Participants) | 50437 | 33415 | 56192 | 40358
Participants | 5404 | 3834 | 6039 | 4458
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - All ED Patients vs Code Sepsis Post-implementation (Intervention Site) - All ED Patients vs Pre-implementation Usual Care (Control Sites) - All ED Patients vs Post-implementation Usual Care (Control Sites) - All ED Patients; Differences-in-differences analysis using multivariable logistic regression to estimate the change in outcome after versus before intervention implementation at the intervention site adjusted for the change observed at control sites and for prespecified covariates; Test type: Superiority — Multiple imputation was employed to account for missing covariate data affecting 3.6% of eligible patients; p = 0.005, Regression, Logistic — Model adjusted for age, sex, Elixhauser Comorbidity Score, ED arrival via ambulance, language preference, temperature, systolic blood pressure, Acute Physiology Score, Sequential Organ Failure Assessment score, and ED-diagnosed source of infection; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.03 to 1.17] — Change in antimicrobial treatment risk associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

8. Other Pre Specified Outcome: Adverse Effects of Antibiotics (Sepsis Patients)
Description: Measured as the fraction of sepsis patients with a discharge diagnosis code consistent with anaphylaxis or with an adverse reaction to antibiotics
Time Frame: From the time of ED arrival to hospital discharge (up to 1 year, average 14 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2384 | 2075 | 2976 | 2716
Participants | 79 | 66 | 79 | 63
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.73, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.68 to 1.75] — Change in risk for possible antimicrobial-associated adverse event associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

9. Other Pre Specified Outcome: Adverse Effect of Antibiotics (All ED Patients)
Description: Measured as the fraction of all ED patients with a discharge diagnosis code consistent with anaphylaxis or with an adverse reaction to antibiotics
Time Frame: From the time of ED arrival to hospital discharge (up to 1 year, average 14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - All ED Patients | Code Sepsis Post-implementation (Intervention Site) - All ED Patients | Pre-implementation Usual Care (Control Sites) - All ED Patients | Post-implementation Usual Care (Control Sites) - All ED Patients
Number analyzed (Participants) | 50437 | 33415 | 56192 | 40358
Participants | 259 | 172 | 287 | 202
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - All ED Patients vs Code Sepsis Post-implementation (Intervention Site) - All ED Patients vs Pre-implementation Usual Care (Control Sites) - All ED Patients vs Post-implementation Usual Care (Control Sites) - All ED Patients; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Multiple imputation was employed to account for missing covariate data affecting 3.6% of eligible patients; p = 0.90, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.78 to 1.33]; Change in risk for possible antimicrobial-associated adverse event associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

10. Other Pre Specified Outcome: New Onset Clostridium Difficile Colitis Incidence (Sepsis Patients)
Description: Incidence of positive stool test for Clostridium difficile colitis between 72 hours and 90 days after ED arrival among ED sepsis patients and (2) all ED patients.
Time Frame: Beginning 72 hours after ED arrival to 90 days after ED arrival
Population: Restricted to participants who met sepsis criteria (acute organ failure plus suspected or confirmed infection) before ED departure. Patients with a positive stool test for Clostridium difficile colitis at baseline (from 14 days prior to ED arrival to 72 hours after ED arrival) were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2354 | 2054 | 2944 | 2686
Participants | 28 | 20 | 44 | 30
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.94, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.49 to 2.17] — Change in new-onset Clostridium difficile colitis risk associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

11. Other Pre Specified Outcome: New Onset Clostridium Difficile Colitis Incidence (All ED Patients)
Description: Incidence of positive stool test for Clostridium difficile colitis between 72 hours and 90 days after ED arrival among all ED patients.
Time Frame: Beginning 72 hours after ED arrival to 90 days after ED arrival.
Population: Patients with a positive stool test for Clostridium difficile colitis at baseline (from 14 days prior to ED arrival to 72 hours after ED arrival) were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-implementation Usual Care (Intervention Site) - All ED Patients | Code Sepsis Post-implementation (Intervention Site) - All ED Patients | Pre-implementation Usual Care (Control Sites) - All ED Patients | Post-implementation Usual Care (Control Sites) - All ED Patients
Number analyzed (Participants) | 50363 | 33376 | 56088 | 40288
Participants | 104 | 61 | 172 | 79
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - All ED Patients vs Code Sepsis Post-implementation (Intervention Site) - All ED Patients vs Pre-implementation Usual Care (Control Sites) - All ED Patients vs Post-implementation Usual Care (Control Sites) - All ED Patients; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Multiple imputation was employed to account for missing covariate data affecting 3.6% of eligible patients; p = 0.10, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.93 to 2.14] — [estimate comment as in outcome 10, analysis 1]

12. Other Pre Specified Outcome: Antibiotic Overtreatment Rate
Description: Fraction of ED patients with a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection who received antibiotics in the ED
Time Frame: Up to 24 hours from ED arrival (an average of 6 hours)
Population: Restricted to patients who had a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection
Measure: Count of Participants; unit: Participants
Groups:
- Pre-implementation Usual Care (Intervention Site) - Sepsis Mimic Patients: Adult patients age ≥18 years who had a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection and who received usual care after presenting to the intervention hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation).
- Code Sepsis Post-implementation (Intervention Site) - Sepsis Mimic Patients: Adult patients age ≥18 years who had a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection and who presented to the intervention hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation).
  Code Sepsis protocol (full implementation): Implementation of a coordinated, structured, multidisciplinary team-based protocol for initial evaluation and treatment of ED patients with suspected sepsis.
- Pre-implementation Usual Care (Control Sites) - Sepsis Mimic Patients: Adult patients age ≥18 years who had a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection and who received usual care after presenting to the control hospital emergency department before implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
- Post-implementation Usual Care (Control Sites) - Sepsis Mimic Patients: Adult patients age ≥18 years who had a primary hospital discharge diagnosis of congestive heart failure or venous thromboembolism and no discharge diagnosis consistent with infection and who received usual care after presenting to the control hospital emergency department after implementation of sepsis care reorganization (Code Sepsis implementation) at the intervention hospital.
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Mimic Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Mimic Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Mimic Patients | Post-implementation Usual Care (Control Sites) - Sepsis Mimic Patients
Number analyzed (Participants) | 1073 | 878 | 1081 | 940
Participants | 48 | 42 | 45 | 58
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Mimic Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Mimic Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Mimic Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Mimic Patients; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Multiple imputation was employed to account for missing covariate data affecting 3.1% of eligible patients; p = 0.59, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.69 to 1.93] — Change in risk for antimicrobial administration in the ED associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

13. Other Pre Specified Outcome: Antibiotic Spectrum (Sepsis Patients)
Description: Total antibiotic spectrum score for all unique antibiotics administered in first 24 hours using antibiotic spectrum scoring system developed by Stenehjem et al. (Clin Infect Dis 2016;63:1273-1280). Individual antibiotics have spectrum scores of 1 to 5, with the total score resulting from summation of the spectrum scores for each unique antibiotic administered during the first 24 hours. Minimum total 24-hour score is therefore 1 (administration of a single, minimum-spectrum antibiotic), with no maximum score. Higher values represent treatment with antibiotics with a broader spectrum.
Time Frame: Up to 24 hours from ED arrival (an average of 6 hours)
Population: Restricted to participants who met sepsis criteria (acute organ failure plus suspected or confirmed infection) before ED departure. Patients who did not receive antibiotics (i.e., received no antimicrobials or received only antivirals or other non-antibiotic classes of antimicrobials) were excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pre-implementation Usual Care (Intervention Site) - Sepsis Patients | Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients | Pre-implementation Usual Care (Control Sites) - Sepsis Patients | Post-implementation Usual Care (Control Sites) - Sepsis Patients
Number analyzed (Participants) | 2337 | 2044 | 2942 | 2704
score on a scale | 5 [3 to 9] | 5 [3 to 9] | 5 [3 to 8] | 4 [3 to 7]
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - Sepsis Patients vs Code Sepsis Post-implementation (Intervention Site) - Sepsis Patients vs Pre-implementation Usual Care (Control Sites) - Sepsis Patients vs Post-implementation Usual Care (Control Sites) - Sepsis Patients; Differences-in-differences analysis using multivariable ??? regression to estimate the change in outcome after versus before intervention implementation at the intervention site adjusted for the change observed at control sites and for subjects' age, sex, Elixhauser Comorbidity Score, ED arrival via ambulance, English language preference, temperature, systolic blood pressure, Acute Physiology Score, Sequential Organ Failure Assessment score, and ED-diagnosed source of infection; Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [0.06 to 0.58] — Change in total spectrum score of antibiotics administered within 24 hours of ED arrival associated with Code Sepsis implementation derived from adjusted differences-in-differences analysis

14. Other Pre Specified Outcome: Antibiotic Spectrum (All ED Patients)
Description: as for outcome 13
Time Frame: Up to 24 hours from ED arrival (an average of 6 hours)
Population: Patients who did not receive antibiotics (i.e., received no antimicrobials or received only antivirals or other non-antibiotic classes of antimicrobials) were excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pre-implementation Usual Care (Intervention Site) - All ED Patients | Code Sepsis Post-implementation (Intervention Site) - All ED Patients | Pre-implementation Usual Care (Control Sites) - All ED Patients | Post-implementation Usual Care (Control Sites) - All ED Patients
Number analyzed (Participants) | 6379 | 4672 | 7634 | 5826
score on a scale | 3 [3 to 5] | 3 [3 to 5] | 3 [3 to 5] | 3 [3 to 5]
Statistical Analysis 1: Comparison: Pre-implementation Usual Care (Intervention Site) - All ED Patients vs Code Sepsis Post-implementation (Intervention Site) - All ED Patients vs Pre-implementation Usual Care (Control Sites) - All ED Patients vs Post-implementation Usual Care (Control Sites) - All ED Patients; Differences-in-differences analysis using multivariable linear regression to estimate the change in outcome after versus before intervention implementation at the intervention site adjusted for the change observed at control sites and for prespecified covariates; Test type: Superiority — Multiple imputation was employed to account for missing covariate data affecting 2.0% of eligible patients; p = 0.02, Regression, Linear; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.03 to 0.31] — [estimate comment as in outcome 13, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Reportable adverse events of anaphylaxis or anaphylaxis-like adverse events were defined as events occurring within 72 hours of ED arrival in the subset of subjects who met sepsis criterial in the emergency department. Per protocol, reportable serious adverse events and non-serious adverse events were defined as events possibly, probably, or definitely related to study procedures (or of uncertain relationship). Non-reportable serious and non-serious adverse events were not recorded.
Arm/Group | Pre-implementation Usual Care (Intervention Site) | Code Sepsis Post-implementation (Intervention Site) | Pre-implementation Usual Care (Control Sites) | Post-implementation Usual Care (Control Sites)
All-Cause Mortality (participants affected / at risk) | 2085/50437 | 1426/33415 | 2520/56192 | 1760/40358
Serious Adverse Events (participants affected / at risk) | 0/50437 | 0/33415 | 0/56192 | 0/40358
Other Adverse Events (participants affected / at risk) | 2/50437 | 3/33415 | 1/56192 | 2/40358
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pre-implementation Usual Care (Intervention Site) (N=50437) | Code Sepsis Post-implementation (Intervention Site) (N=33415) | Pre-implementation Usual Care (Control Sites) (N=56192) | Post-implementation Usual Care (Control Sites) (N=40358)
Anaphylaxis (Immune system disorders) | 2/2384 | 3/2075 | 1/2976 | 2/2716 — Anaphylaxis or anaphylaxis-like clinical event occurring within 72 hours of hospital arrival among patients meeting sepsis criteria before emergency department departure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT04148989/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT04148989/SAP_001.pdf